CLINICAL TRIAL: NCT03914430
Title: The Effect of Dairy and Non-Dairy Cultured Products Added to Breakfast Cereals on Satiation, Satiety, Blood Glucose Control and Short-Term Food Intake in Young Adults
Brief Title: Breakfast Cereals Consumed in Dairy and Non-dairy Medium: the Effects on Blood Glucose, Satiety and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Collaborators: University of Toronto (Other); Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Bohdan Luhovyy, Associate Professor, Mount Saint Vincent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2015-013
Record Dates: First submitted 2019-04-02; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Blood Glucose; Eating; Food
Keywords: Breakfast; Blood glucose; Food intake; Satiety
MeSH Terms: interventions — Food

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants were blinded and could not distinguish the breakfast cereals made with Greek yogurt or with cultured coconut product. The taste and flavour in both treatments was similar due to added blueberry flavouring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breakfast meal with granola cereal and cultured dairy (Experimental)
  Interventions: Other: Food
- Breakfast meal with granola cereal and cultured non-dairy (Experimental)
  Interventions: Other: Food
- Water (Experimental): Energy-free control
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — The intervention represents a breakfast meal (cereals with cultured products) or breakfast skipping (water control)

SUMMARY:
The effects of dairy-free products consumed with a breakfast meal on food intake and glycaemic regulation remain unexplored. It is known that dairy products are an excellent source of protein, low glycaemic sugar lactose, calcium, and vitamin D. In our recent study the consumption of a dairy snack with high protein content resulted in reduced blood glucose response compared to non-dairy snack with the similar amount of available carbohydrate. The investigators hypothesize that the ad libitum intake of breakfast cereals served with a high-protein fermented dairy product will result in reduced and sustained blood glucose response compared to non-dairy control. The objective of this study is to investigate how dairy and non-dairy cultured products used as carriers for breakfast granola cereals and consumed ad libitum affect short-term food intake, satiety, and glycaemia within two hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females

Exclusion Criteria:

* Overweight or obese
* Breakfast skippers
* Have any chronic metabolic diseases
* Smokers
* Taking medications

Ages: 19 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose concentration | 0-120 minutes
  The concentration of blood glucose in venous blood after the ad libitum breakfast meal or water control.
Subjective feeling of appetite | 0-120 minutes
  The subjective assessment of appetite parameters including desire to eat, fullness, hunger and a prospectiove food consumption measured with 100 mm Visual Analogue Scales with two opposite statements at each end (e.g., for the hunger scale, 0 mm means not hungry at all, and 100 mm means very hungry).
Ad libitum food intake | 0-120 minutes
  The amount of energy (kcal) consumed ad libitum with the breakfast meal or water control and with the test meal (pizza lunch) two hour later.

SECONDARY OUTCOMES:
Circulatory insulin concentration | 0-120 minutes
  The concentration of insulin in blood
Subjective feeling of physical comfort | 0-120 minutes
  The subjective assessment of wellness and gastrointestinal symptoms including feeling of nausea, diarrhoea, flatulence and other parameters measured with 100 mm Visual Analogue Scales with two opposite statements at each end.
Subjective feeling of food palatability (pleasantness) | 0, 120 minutes
  The pleasantness of the breakfast meal and pizza meal measured with 100 mm Visual Analogue Scales with two opposite statements at each end.(e.g., 0 mm means that food is not pleasant at all, and 100 mm means that the food is very pleasant).

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Luhovyy, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No